CLINICAL TRIAL: NCT04053517
Title: Frequency and Correlates of Financial Distress in Advanced Cancer Patients
Brief Title: Financial Distress in Advanced Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0694; NCI-2019-03869 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0694 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-07-15; First posted 2019-08-12 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Neoplasm; Locally Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm; Refractory Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire administration): Patients complete questionnaires about financial state and quality of life over 15 minutes. Patients' medical chart is also reviewed.
  Interventions: Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Medical Chart Review — Medical chart is reviewed
  Other Names: Chart Review
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the severity of financial distress in advanced cancer patients. The cost of cancer care can often be very expensive. Financial distress from the burdens of high costs and debt may interfere with a patient's physical symptoms and quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the frequency of high financial distress in advanced cancer patients.

SECONDARY OBJECTIVES:

I. To determine the association between high financial distress with clinical and demographic characteristics in advanced cancer patients.

II. To determine the correlation between In Charge Financial Distress/ Financial Well-Being Scale (IFDFW) and other financial distress instruments such as Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT) and Edmonton Symptom Assessment Scale- Financial Distress (ESAS-FS).

III. To determine the association between high financial distress with patient symptoms in ESAS-FS and quality of life assessed by the Functional Assessment of Cancer Therapy - General (FACT-G).

OUTLINE:

Patients complete questionnaires about financial state and quality of life over 15 minutes. Patients' medical chart is also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosis of advanced cancer, as defined by recurrent disease, locally advanced disease, metastatic disease, or refractory disease
* Patients must be able to understand, read, write, and speak English
* Patients must have no clinical evidence of severe cognitive impairment (Memorial Delirium Assessment Scale score of >= 13) and should be able to consent and answer the questionnaires
* Patients must sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of advanced cancer
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
InCharge Financial Distress/Financial Well-Being Scale (IFDFW), | Day 1
  a validated survey designed to measure a person's financial state, consists of eight questions and each of them is rated from 1 (overwhelming stress) to 10 (no stress at all). This should take approximately 5 minutes to complete.

SECONDARY OUTCOMES:
Correlation between high financial distress with clinical characteristics in advance cancer patients | Day 1
  Demographic and clinical characteristics,such as your age, gender, ethnicity, caregiving, education, employment status, marital status, household income, date of diagnosis, disease stage, cancer type, insurance type, place of residence, and homeowner status) will be collected. It should take about 5 minutes to complete.
Correlation between mean scores of In Charge Financial Distress/ Financial Well-Being Scale (IFDFW) and scores from other financial distress instruments | Day 1
  Comprehensive Score for Financial Toxicity Functional Assessment of Chronic Illness Therapy (COST-FACIT) was developed as part of a series of questionnaires aimed at measuring different symptom indexes of health-related quality of life in patients with advance disease such as cancer. The survey contains 12 questions and each of them is rated from 0 (not at all) to 4 (very much). This survey focuses on financial distress caused by illness in patients with cancer. It takes about 5 minutes to complete.
Correlation between high financial distress with patient symptoms in(ESAS) Edmonton Symptom Assessment System | Day 1
  Edmonton Symptom Assessment Scale- Financial Distress (ESAS-FS) is routinely utilized in the outpatient Supportive Care Clinic. The ESAS-FS is an updated version including financial and spiritual distress, and it consists of 12 symptom items to measure severity severity of patient's symptoms. Grading severity of patient symptoms from "no" 0 to "worst symptom" 10 in the last 24 hours.
Correlation between high financial distress with Quality of life | Day 1
  Functional Assessment of Cancer Therapy - General (FACT-G). consists of 27 general questions divided into four primary domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being for use in patients with any form of cancer. Answered using a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much) With a total possible score greater than 100.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Tschanz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org